CLINICAL TRIAL: NCT00295178
Title: A Multicenter, Randomized Study Comparing CUBICIN® (Daptomycin for Injection) With Vancomycin in the Treatment of Cellulitis or Erysipelas
Brief Title: Study Comparing CUBICIN® (Daptomycin for Injection) With Vancomycin in Cellulitis or Erysipelas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3009-008; DAP-4CELL-05-02 (Other: Cubist)
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Cellulitis
MeSH Terms: conditions — Cellulitis | interventions — Daptomycin; Vancomycin

INTERVENTIONS:
Drug: Daptomycin
Drug: Vancomycin

SUMMARY:
This study is designed to investigate the difference in speed and degree of symptom resolution between daptomycin and vancomycin in subjects treated for cellulitis or erysipelas by evaluation of the following parameters:

* Time to erythema margin cessation to progress
* Time to defervescence
* Time to hospital discharge following relief of the presenting cellulitis or erysipelas
* Degree of improvement of the following signs and symptom of cellulitis or erysipelas including
* Degree of improvement of cellulitis-related pain and swelling as reported by subjects

Additionally, the difference in frequency of Adverse Events between daptomycin and vancomycin will be described.

DETAILED DESCRIPTION:
same as above

ELIGIBILITY:
Inclusion Criteria:

1. Read and sign the informed consent form after the nature of the study has been fully explained;
2. Male or female > or = 18 years of age;
3. If female of childbearing potential, a negative pregnancy test is required;
4. Primary diagnosis of cellulitis/ erysipelas

   1. with onset of signs or symptoms within 3 days of 1st dose of study medication
   2. requiring hospitalization, and severe enough to warrant IV antibiotics
   3. temperature >37.5°C (99.5° F) oral or >38° C (100.2° F) rectal, documented within 48 hours prior to enrollment, and
   4. anticipated treatment to be limited to medical (NOT surgical) interventions
   5. at an anatomical location that allows of a clear assessment of the erythema margin

Exclusion Criteria:

1. Pregnant or lactating female;
2. Conditions where required surgery (in and of itself) constitutes curative treatment of the infection or removal of infected site (e.g., amputation);
3. Conditions requiring emergent surgical intervention at the site of infection (e.g., progressive necrotizing infections);
4. Previous systemic antimicrobial therapy exceeding 24 hours duration, administered anytime during the 72 hours prior to the first dose of study drug unless on previous antibiotics for at least 72 hours and without any clinical improvement;
5. Cellulitis associated with a wound infection or ulcer requiring incision and drainage or debridement
6. Perirectal abscess or hidradenitis suppurativa or third degree burn infections
7. Buccal cellulitis, facial cellulitis, perianal cellulitis, or periorbital cellulitis;
8. Known or suspected osteomyelitis, pneumonia, bacteremia, endocarditis, or urinary tract infection;
9. Known to be allergic or intolerant to study medications;
10. Subjects with a Creatinine Clearance (CLCR) <30 mL/min;
11. Requirement for non-study systemic antibiotics;
12. Requirement for systemic steroids from enrollment through stabilization of cellulitis;
13. Rhabdomyolysis;
14. Neutropenic subjects with absolute neutrophil count ≤ 500 cells/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-02-20 (Actual); Primary Completion 2006-08-09 (Actual); Study Completion 2006-08-09 (Actual)

PRIMARY OUTCOMES:
investigating the differences in speed and degree of symptom resolution between CUBICIN and vancomycin

SECONDARY OUTCOMES:
frequency of Serious Adverse Events between daptomycin and vancomycin will be described

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Friedman, MD, Principal Investigator — Joseph M. Still Research Foundation, Inc.
Locations (1):
- Joseph Still Research Foundation, Augusta, Georgia, United States

REFERENCES:
- [Derived] Pertel PE, Eisenstein BI, Link AS, Donfrid B, Biermann EJ, Bernardo P, Martone WJ. The efficacy and safety of daptomycin vs. vancomycin for the treatment of cellulitis and erysipelas. Int J Clin Pract. 2009 Mar;63(3):368-75. doi: 10.1111/j.1742-1241.2008.01988.x. PMID 19222623